CLINICAL TRIAL: NCT03268200
Title: The Effect of Segmental Re-examination of Colon for Adenoma Detection in Colonoscopy: a Randomized, Controlled Trial
Brief Title: The Effect of Segmental Re-examination of Colon for Adenoma Detection in Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jeong-Seon Ji, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: reexamination
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Adenoma
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): Each segment of colon (right colon, mid-colon, and left colon) was examined twice
  Interventions: Other: segmental reexamination
- Control group (No Intervention): Withdrawal time in the each segment of colon (right colon, mid-colon, and left colon) was about 2 minutes.

INTERVENTIONS:
Other: segmental reexamination — segmental reexamination during colonoscopy
  Arms: Case group

SUMMARY:
The aim of this study was to determine whether segmental re-examination of the each segment (right colon, mid-colon, and left colon) could increase the proximal adenoma detection rate (ADR) and to evaluate the time-effectiveness of this approach.

DETAILED DESCRIPTION:
The investigators prospectively recruited patients (aged ≥45 and ≤75 years) who were scheduled to undergo colonoscopy at our center. Patients were excluded if they had advanced colonic cancer, prior resection of the proximal colon, inflammatory bowel disease, or polyposis syndrome, or were unable to provide informed consent. In addition, if the quality of bowel preparation was unsatisfactory (Boston Bowel Preparation Scale [BBPS] score <2 in any segment of the colon), or if the cecum could not be intubated during the colonoscopy, patients were excluded.

A randomization list was generated with the randomization algorithm of random sorting, using Excel program. Included patients were randomly assigned to one of the two groups: segmental re-examination group, in which the each segment (right colon, mid-colon, and left colon) was examined twice segmentally; or control group, in which the withdrawal time in the each segment was about 2 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients (aged ≥45 and ≤75 years) who were scheduled to un- dergo colonoscopy

Exclusion Criteria:

* Patients who had advanced colonic cancer, prior resection of the proximal colon, inflammatory bowel disease, or polyposis syndrome, or were unable to provide informed consent.
* If the quality of bowel preparation was unsatisfactory (Boston Bowel Preparation Scale [BBPS] score <2 in any segment of the colon), or if the cecum could not be intubated during the colonoscopy, patients were excluded.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 7 days

SECONDARY OUTCOMES:
Per-patient adenoma detection rate (ADR) at each segment of colon | 7 days
per-patient polyp detection rate | 7 days
Withdrawal time | 1 days

CONTACTS AND LOCATIONS:
Locations (1):
- Incheon St. Mary's hospital, Catholic university of Korea, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee DS, Ji JS, Gweon TG, Seo M, Choi H. Efficacy of colonoscopic re-examination across the entire colon: a randomized controlled trial. Surg Endosc. 2024 Nov;38(11):6711-6717. doi: 10.1007/s00464-024-11298-5. Epub 2024 Sep 26. PMID 39327294